CLINICAL TRIAL: NCT00468780
Title: Study to Evaluate the Safety and Efficacy of Redirecting Ambulance Patients to Destinations Based on Acuity
Brief Title: Standardized Comparison of Triage in EMS
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 724180022
Record Dates: First submitted 2007-05-01; First posted 2007-05-03 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
Keywords: Canadian Triage Acuity Scale; paramedics; triage nurse; triage levels; inter-rater reliability; health services outcomes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to evaluate the reliability and validity of acuity estimates by paramedics employing the Canadian Triage Acuity Scale (CTAS) in the out of hospital setting. The study has the potential to help guide policy decisions pertaining to the safe transfer of ambulance patients to alternative destinations reducing ED overcrowding and ambulance off load time. Emergency Department triage nurses employ the same acuity scale and if this study is successful the emergency departments and the EMS services could communicate about capacity to handle patients based on acuity, volumes and waiting times.

DETAILED DESCRIPTION:
CTAS stands for the Canadian Triage Acuity Scale. CTAS defines 5 levels of triage according to the perceived need for physician assessment. CTAS was developed to measure ED case mix and evaluate the potential effect of changes in the delivery of health care on patients seeking emergency care. Although the Canadian Institute of Health Information (CIHI) collects data on total visits, admissions, and ambulatory care visits, there are few standards for reporting data from Emergency Departments. The Canadian Association of Emergency Physicians endorsed CTAS as a standardized data element to assess and compare case mix and acuity.

At present there are no consistently utilized measures of patient acuity performed by paramedics in Ontario. Information on the interface between Prehospital Care and Emergency Departments would inform decision-making on the Emergency Health Care system. The introduction of CTAS provides a superb opportunity to evaluate its utility in providing this information on an accurate and consistent basis.

The use of an acuity scale common to the in-hospital and prehospital setting seems ideal. However, there are several questions to be answered regarding the feasibility, reliability, safety and validity of CTAS before widespread implementation. The Society for Academic Emergency Medicine's position clearly states, "Patients may be referred to other locations where they will receive care appropriate to the acuity of their problem only if the triage criteria, if any, are based on research that shows them to be safe and effective". In their prospective trial, Brillman et al. noted that 26-38% of emergency department patients who were admitted to hospital would not have been identified at triage even when the treating physician assessed them. If physicians are not capable of accurate triage decisions, one must consider the reliability of a paramedic under the challenges of the prehospital setting. Moreover, recent high-profile coroner cases suggest that liability is a significant concern. Paramedics are accustomed to point-of-care assessment and triage, and do not have access to some of the resources utilized by ED nurses. Because the environment, context, discriminating tools, resources and skill set differ between triage nurses and paramedics, it is essential to evaluate the use of paramedic assessment tools in the determination of an accurate and consistent CTAS score. Moreover there has not as yet been an emphasis on paramedic assessment interfacing with decision-making and time to care. It is important to ensure, therefore, that the prehospital application of CTAS is appropriate and safe.

The objectives of this study are to evaluate the criterion validity of CTAS assignment by paramedics at departure from scene and arrival at hospital compared to a CTAS expert (gold standard), to evaluate the inter-rater reliability of CTAS assignment by paramedics at arrival at hospital compared to triage nurses, to evaluate the predictive validity of CTAS level assignment with respect to patient outcomes and health care resource utilization and to describe the relationship and the use of the return priority code and the CTAS category.

A random sample of Advanced Care Paramedic crews and an equal number of randomly selected Basic Care Paramedic crews from five EMS systems (rural and urban) will be invited to participate. A paramedic observer (advanced and basic) with advanced CTAS skills will observe each crew, record the critical elements of each prehospital encounter on a data collection sheet and assign a CTAS level to the patient on departure from scene and arrival at hospital. The observer will also record the CTAS level and return priority code conveyed by the paramedic to the dispatch centre, and evaluate whether the use of both the return priority code (in which an urgent return is assigned a value of 4) and the CTAS score (in which an urgent call is assigned a value of 1 or 2) generates any difficulties in paramedic communication with dispatch on departure from the scene.

At the hospital, the observer will ensure that the triage nurse assigns the CTAS level without prior knowledge of the paramedic assignment. The observer will record the CTAS level assigned by the triage nurse as well as the CTAS level at departure from the scene and on arrival at the receiving hospital, return priority code and status change code recorded by the treating paramedic on the ambulance call report. The patient's health insurance number (HIN) will be collected for the purposes of linkage to outcome data. The observer will record the times of departure from scene and arrival at hospital to estimate the transport interval.

Validity will be measured by calculating a kappa statistic comparing the observer's (gold standard) CTAS score with the paramedic CTAS score at departure from scene and arrival at hospital.

Inter-rater reliability of CTAS between medics (as assigned at arrival at hospital) and triage nurses will be estimated using a kappa statistic. The same measure of agreement will be estimated between the triage nurse and the observer.

Agreement between the return priority code initially conveyed by the paramedic to dispatch and the code recorded on the ACR will be evaluated using the kappa statistic. The relationship between CTAS score and return priority code will be measured using descriptive statistics and non-parametric correlation. The frequency of calls in which problems in paramedic communication with dispatch arose with respect to the use of both CTAS and return priority will be calculated and the types of problems encountered described.

ELIGIBILITY:
Inclusion Criteria:

* All patients

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study is taking place in 7 EMS systems in Ontario: Peterborough, Thunder Bay, Hamilton, Simcoe/Muskoka, Durham, Peel, and Toronto.
  The participants(Both Primary care paramedics and Advance Care Parmaeidcs)are riding as civilian observers under contract to the Sunnybrook and Women's College Health Sciences Centre Research Institute and have signed liability release forms.
  The main focus of the SCORE study is to determine how well paramedics in the field can correctly assign CTAS scores. By showing that it can be done reliably, decisions can be made on suitable destinations, especially for the low acuity patient.
Sampling Method: Probability Sample
Enrollment: 928 (Actual)
Dates: Start 2003-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
CTAS level assignment | At the time of departue from scene and arrival at hospital
  Reliability and validity of CTAS level assignment by paramedics and EMS service implementation

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Morrison, MD, Principal Investigator — Sunnybrook Health Sciences Center
Locations (2):
- Canada (2):
  - Hamilton Health Sciences, Hamilton, Ontario
  - Sunnybrook-Osler Centre for Prehospital Care, Toronto, Ontario